CLINICAL TRIAL: NCT06515093
Title: A Randomized Post-Market Study Assessing Complete Wound Healing by Comparing Surgenex® PelloGraft in Treating Diabetic Foot Ulcers (DFU) and SanoGraft® in Treating Venous Leg Ulcers (VLU) to SOC Treatment
Brief Title: Study Assessing Complete Wound Healing by Comparing Surgenex® PelloGraft in Treating DFU and SanoGraft® in Treating VLU to SOC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Surgenex (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-SUR-001
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-08

CONDITIONS: Diabetic Foot Ulcer; Venous Leg Ulcer
MeSH Terms: conditions — Diabetic Foot; Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 PelloGraft (Experimental): PelloGraft treatment for diabetic foot ulcers versus Standard of Care treatment for diabetic foot ulcers
  Interventions: Other: PelloGraft
- Arm 2 SanoGraft (Experimental): SanoGraft treatment for venous leg ulcers vs Standard of Care treatment for venous leg ulcers
  Interventions: Other: SanoGraft

INTERVENTIONS:
Other: PelloGraft — dual layer amnion/chorion-derived allograft
  Arms: Arm 1 PelloGraft
Other: SanoGraft — single layer amnion-derived allograft
  Arms: Arm 2 SanoGraft

SUMMARY:
The purpose of this study is to compare Pellograft to standard of care modalities in treating diabetic foot ulcers in human subjects, and to compare Sanograft to standard of care in treating venous leg ulcers. The study will demonstrate wound healing outcomes with comparators including time to wound epithelialization, decrease in wound size, and total number of study product applications towards healing outcome. This information is important to the Centers for Medicare and Medicaid Services (CMS) and other payors in determining coverage policy and reimbursement for this product category.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years of age
2. Diabetic Foot Ulcer Only - Subject has diagnosed Type 1 or Type 2 diabetes
3. Subject's wound is located on foot or ankle (DFU) or leg (VLU)
4. Subject has diabetic foot ulcer > 1.0 cm2 and ≤ 25 cm2 OR venous leg ulcer > 1.0 cm2 and ≤ 50 cm2
5. Subject has adequate circulation to affected extremity with TcPO2 results of ≥ 40 mm Hg on the dorsum of the affected foot or ABI results ≥ 0.7 and≤ 1.2 or Great Toe Pressure ≥ 50 mmHg
6. Subject is willing and able to comply with all protocol requirements
7. Subject is willing and able to provide informed consent or obtain consent from legal authorized representative (LAR)

Exclusion Criteria:

1. Subject is pregnant
2. Subject with diagnosed diabetes has HbA1C > 12 within 3 months Prior to randomization
3. Subject has > 30% reduction in wound size after 2-week run-in period
4. Subject has active infection, undrained abscess, or critical colonization of the wound with bacteria
5. Subject has osteomyelitis or joint capsule on investigator's exam or radiographic evidence or bone culture, histology, x-ray changes or MRI
6. Subject is on parenteral corticosteroids or any cytotoxic agents for 7 consecutive days during 30 days before screening. Chronic oral steroid use is not excluded if dose < 10 mg per day of prednisone
7. Subject is currently undergoing cancer treatment
8. Subject has used biologic skin substitutes within 14 days of enrollment
9. Subject has an allergy to suture material
10. Subject has life expectancy less than six-months as assessed by the investigator
11. Subject is participating in another clinical research study prior to this study completion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-06-23 (Actual); Primary Completion 2026-03-26 (Estimated); Study Completion 2026-09-09 (Estimated)

PRIMARY OUTCOMES:
100% epithelialization | 12 weeks (DFU) or 16 weeks (VLU)
  100% epithelialization of wound within 12 weeks (DFU) or 16 weeks (VLU) of initial treatment application. Wound closure is complete with confirmation of 100% epithelialization, no drainage, and no need for additional dressings.

SECONDARY OUTCOMES:
Time to Healing | 12 weeks (DFU) or 16 weeks (VLU)
  Time to Healing (from initial application of study product to 100% epithelialization of wound)

OTHER OUTCOMES:
Quality of Life via subject questionnaire | 2-weeks post wound closure
  Qualify of Life at 2-week post closure follow-up via SF-36 Questionnaire

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - ILD Research, Vista, California
  - Future Life Clinical Trials, North Miami, Florida
  - Boston Medical Center, Boston, Massachusetts
  - Essential Medical Research, Tulsa, Oklahoma